CLINICAL TRIAL: NCT03592069
Title: 10 Day Concomitant Versus 14 Day Hybrid Regimen as First Line H. Pylori Eradication Treatment in a High Clarithromycin Resistance Area. A Multicenter Randomized Equivalence Trial
Brief Title: Concomitant Versus Hybrid Regimen for H. Pylori Eradication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandra Hospital, Athens, Greece (Other)
Collaborators: Hellenic Society of Gastroenterology (Unknown)
Responsible Party: Principal Investigator, SPYRIDON MICHOPOULOS, Head of GI Department, PhD, MD, Alexandra Hospital, Athens, Greece
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlexandraH
Record Dates: First submitted 2018-06-13; First posted 2018-07-19 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: H.Pylori Infection; H.Pylori Gastrointestinal Disease; H. Pylori Associated Phlegmonous Gastritis
Keywords: H. Pylori Infection; Gastritis; H.Pylori treatment; Treatment Resistance
MeSH Terms: conditions — Gastritis | interventions — Clarithromycin; Metronidazole; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 day concomitant (Active Comparator): After the confirmation of H. pylori infection, eligible patients randomly assigned to either concomitant or hybrid treatment group will receive:
  - Concomitant for 10 days, including 40 mg of esomeprazole bid, amoxicillin 1g bid, clarithromycin 500mg bid and metronidazole 500mg bid.
  Interventions: Drug: 10 day concomitant regimen
- 14 day hybrid (Active Comparator): After the confirmation of H. pylori infection, eligible patients randomly assigned to either concomitant or hybrid treatment group will receive:
  Hybrid for 14 days, including 40 mg of esomeprazole bid and amoxicillin 1g bid, for the first 7 days followed by esomeprazole 40mg bid, amoxicillin 1g bid, clarithromycin 500mg bid and metronidazole 500mg bid, for another 7 days.
  Interventions: Drug: 14 day hybrid regimen

INTERVENTIONS:
Drug: 10 day concomitant regimen — 10 Day Concomitant Hp therapy Concomitant for 10 days, including 40 mg of esomeprazole bid, amoxicillin 1g bid, clarithromycin 500mg bid and metronidazole 500mg bid
  Other Names: Amoxicillin 1gr bid from day 1 to day 10; Clarithromycin 500mg bid from day 1 to day 10; Metronidazole 500mg bid from day 1 to day 10; Esomeprazole 40mg bid from day 1 to day 10
  Arms: 10 day concomitant
Drug: 14 day hybrid regimen — 14 Day Hybrid Hp therapy Hybrid for 14 days, including 40 mg of esomeprazole bid and amoxicillin 1g bid, for the first 7 days followed by esomeprazole 40mg bid, amoxicillin 1g bid, clarithromycin 500mg bid and metronidazole 500mg bid, for another 7 days.
  Other Names: Amoxicillin 1gr bid from day 1 to day to day 14; Clarithromycin 500mg bid from day 8 to day 14; Metronidazole 500mg bid from day 8 to day 14; Esomeprazole 40mg bidfrom day 1 to day to day 14
  Arms: 14 day hybrid

SUMMARY:
10 day concomitant versus 14 day hybrid regimen as first line H. pylori eradication treatment in a high clarithromycin resistance area. A multicenter, randomized, equivalence trial.

DETAILED DESCRIPTION:
RESEARCH PROTOCOL:

TITLE "10 day concomitant versus 14 day hybrid regimen as first line H. pylori eradication treatment in a high clarithromycin resistance area. A multicenter, randomized, equivalence trial."

INTRODUCTION

Helicobacter pylori (H. pylori) is a global human pathogen implicated in the pathogenesis of prevalent and serious diseases mainly peptic ulcer disease and gastric malignancy.1 Recent guidelines propose H. pylori eradication every time that it is found with the usual detection methods.2 Successful eradication largely depends on the choice of antibiotics in which the microbe is mostly sensitive.3 Usual first line therapies contained a proton pump inhibitor (PPI) and two antibiotics, clarithromycin with amoxicillin or metronidazole when amoxicillin wasn't indicated.4 Eradication rates have been initially acceptable reaching over 80% in per protocol analyses.5,6 However in late years H. pylori has developed an increasingly high resistance profile which has reached over 20% in most European countries, including ours. As a consequence, eradication rates with triple regimens declined to percentages less than 80% in per protocol analyses.7-9 Currently acceptable schemes include the already known bismouth containing quadruple regimen and the non bismouth quadruples namely concomitant, sequential and hybrid.10,11 In our country the 10 days concomitant regimen presents stable and high eradication rates which are significantly better than the standard triple and sequential regimens of the same duration.12-14 In two recent studies concomitant had a significant advantage over sequential on metronidazole resistant strains as well as on dual resistant to both clarithromycin and metronidazole strains.14,15 The hybrid regimen is the less studied first line regimen in Europe.16 In a recent study, on a Greek population, a 14 days hybrid regimen achieved encouraging results and the only predictive factor for failure has been dual resistance.17 To date there hasn't been any comparative study between 10 days concomitant and 14 days hybrid regimens.16

PURPOSE OF STUDY The investigators designed an equivalence trial between the 10 days concomitant and 14 days hybrid regimens in a Greek population.The investigators primary outcome is to compare total eradication rates between these two regimens in intention to treat and per protocol analyses. Secondary outcomes are to compare eradication rates in respect to genotypic and phenotypic resistance profiles, the effect of antibiotic resistance on therapy, patient's compliance, adverse events and economic evaluation of the two regimens.

PATIENTS - METHODS

Patient selection Patients of 18 years or older with dyspepsia / or iron deficiency anaemia, referring for upper GI endoscopy and found to be infected with H. pylori (positive rapid urease test), naïve to H. pylori eradication treatment, will be invited to participate in the study. Exclusion criteria are: age below 18 years, presence of severe co-morbidities (i.e. liver cirrhosis, renal failure, haematological, neurological, psychiatric, cardiovascular or pulmonary disease), previous gastric surgery, gastric malignancies, Zollinger-Elisson syndrome, known allergy or other contraindications to the study medications, previous H. pylori treatment, use of antibiotics , bismuth salts , NSAIDS or aspirin in the preceding month, use of PPI in the preceding two weeks and not willing to participate in the study. Pregnant or lactating women will also be excluded.

Study Design The study will be prospective. Upper GI endoscopy including two antral biopsies for rapid urease test (CLO-test) will be performed at each patient. In patients tested positive two additional specimens (from the antrum and corpus) will be sent to a reference laboratory for culture and antibiotic susceptibility tests. In cases with indication for histology or equivocal CLO-test results, at least two specimens will be taken from the antrum and corpus respectively, to confirm H. pylori gastritis using haematoxylin-eosin and modified Giemsa staining. In equivocal cases an immunohistochemical method can be used. Patients tested positive by urease test and/or histology will be allocated to either treatment group. Every patient will sign an informed consent in order to participate in the study. Additionally, a careful medical history will be obtained and complete clinical examination performed (including appropriate blood or other tests if indicated) prior to inclusion into the study.

Participants will be randomly assigned, in a 1:1 basis, to one of two treatment groups namely concomitant and hybrid. Randomization will be organized centrally by an independent assistant investigator using a computer-generated randomization method, using a block size of four. This will produce a separate number for each patient sealed in an opaque envelope and kept in his office throughout the study. After obtaining informed consent, the investigators would call the research assistant to open the envelope for the allocated regimen. All data will be inserted in a computer database and elaborated by the participating investigators. The trial is not blinded for patients and recruiting physicians, regarding treatment regimen, as in most randomized controlled H. pylori eradication trials.

Interventions

After the confirmation of H. pylori infection, eligible patients randomly assigned to either concomitant or hybrid treatment group will receive:

* Concomitant for 10 days, including 40 mg of esomeprazole bid, amoxicillin 1g bid, clarithromycin 500mg bid and metronidazole 500mg bid.
* Or Hybrid for 14 days, including 40 mg of esomeprazole bid and amoxicillin 1g bid, for the first 7 days followed by esomeprazole 40mg bid, amoxicillin 1g bid, clarithromycin 500mg bid and metronidazole 500mg bid, for another 7 days.

Esomeprazole will be given before and antibiotics after meals, in both regimens. In the post-treatment period, symptomatic patients will be allowed to use antacids on demand. Antibiotics or other medications interfering with the treatment results will be prohibited during the study period. Efficacy of treatment will be evaluated 4-6 weeks after completion of antibiotic therapy by 13C-urea breath test (13C-UBT) performed according to the standard European protocol. In patients requiring a follow-up endoscopy due to peptic ulcer disease, persisting or recurring symptoms, the diagnostic test of choice will be histological examination of four samples taken, in pairs, from the antrum and from the corpus and stained by modified Giemsa.

Tolerability and adherence Side effects of treatment will be assessed on a structured clinical interview with a specific questionnaire completed immediately after the end of eradication therapy and at the final re-evaluation. During the interview, patients will be asked to grade the severity of each adverse event experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with common everyday activities), or "severe" (causing considerable interference with patients' daily activities).18 Incapacitating or life-threatening complications will be classified as serious and will be reported to regulatory agency (National Organization of Medicines). Adherence to treatment will be assessed by providing all patients with a pre-structured printed table with all dosages illustrated, asking to tick each time a pill was consumed and bring it back along with any tablet not consumed, for pill counting. In case of discrepancies found between the structured printed table and residual medication, the latter will be taken into account to evaluate patient's adherence. Poor adherence is defined as <90% of the total medication taken.

Culture and antibiotic susceptibility tests Isolation of clinical H. pylori strains H. pylori clinical strains will be isolated from gastric biopsies. All biopsies will be placed in thioglycollate medium (Oxoid, Basingstoke, UK) and will be sent to the Laboratory of Medical Microbiology (Hellenic Pasteur Institute) for H. pylori isolation within 2-4 hours after endoscopy. Following addition of sterile glass beads, biopsy samples will be vigorously vortexed and 100μl of homogenate will be cultured for up to 7 days, at 37°C under microaerophilic conditions (CampyPak-Plus, Becton-Dickinson, Cockeysville, MD), on Columbia agar plates containing antibiotics (vancomycin 10μg/mL, trimethoprim 10μg/mL, polymyxin B 104 IU/L, amphotericin B 2μg/mL, nalidixic acid 10μg/mL, bacitracin 30μg/mL and fluorocytosine 5μg/mL), supplemented with 8%v/v horse blood and 1% v/v Vitox (Oxoid, Basingstoke, UK). Culture sweeps, as well as individual colonies will be collected and frozen at -80°C, until used.

Antibiotic susceptibility testing Antibiotic susceptibility testing of H. pylori will be performed utilizing E-test strips (BioMerieux, Marcy l'Étoile, France), according to the manufacturer's instructions, on Mueller Hinton agar medium (Beckton Dickinson) supplemented with 10% horse blood. Briefly, agar plates will be freshly prepared and used within 7 days following their preparation. Bacterial inoculum will be prepared from a 1 or 2 day old culture and bacterial suspension will be adjusted to McFarland 3 turbidity (approx. 108 colony forming units-CFU/mL). E-test strips will be applied with sterile forceps to the dried agar surface, following application of the bacterial inoculum and plates will be incubated at 37°C under microaerophilic conditions. Results will be read at 72 hours. MIC clinical breakpoints used to define resistance according to EUCAST will be: clarithromycin (>0.5 mg/L), levofloxacin (>1 mg/L), tetracycline (>1 mg/L), metronidazole (>8 mg/L) and amoxicillin (>0.12 mg/L). To detect genotypic resistance to clarithromycin and levofloxacin a real time PCR will be implemented in cultured H. pylori strains.

Sample size calculation The study is designed to prove or reject equivalence between the two eradication regimens under study namely 10 days concomitant and 14 days hybrid (equivalence trial). Based on the results of previous studies eradication rates over 85% in intention to treat and over 90% in per protocol analyses have been found for both regimens.17 According to international statistical rules (FDA) two regimens are considered equivalent when the confidence intervals of the difference between their eradication rates do not exceed 15%. Using the Monte Carlo (500 X 500 runs) simulation system and taken into account that in the existing Greek studies14-16 eradication rates for hybrid regimen are between 86 and 90% in intention to treat analysis we calculated a sample size of 150 patients in each treatment arm (with a 10% drop out rate) in order to get an 80% power in the study.

Statistical analysis Comparisons of proportions will be done using the chi-square test. Continuous non-parametric data will be compared using the t test. Stepwise multivariate logistic regression analysis will be performed to evaluate factors influencing H. pylori eradication in patients who had a final treatment outcome with either concomitant or hybrid therapy.

ELIGIBILITY:
Inclusion criteria:

* patients of 18 years or older referring for upper GI endoscopy
* infected with H. pylori (verified with 2 out of 3 tests - rapid urease test, histology, culture)
* without previous H. pylori eradication treatment (naïve)

Exclusion criteria are:

* age below 18 years
* presence of severe co-morbidities (i.e. liver cirrhosis, renal failure, haematological, neurological, psychiatric, cardiovascular or pulmonary disease)
* previous gastric surgery
* gastric malignancies
* Zollinger-Elisson syndrome
* known allergy or other contraindications to the study medications
* previous H. pylori treatment
* use of antibiotics , bismuth salts , NSAIDS or aspirin in the preceding month
* use of PPI in the preceding two weeks
* not willing to participate in the study
* pregnant or lactating women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
To compare eradication rates between a 10 day concomitant and a 14 day hybrid regimens in intention to treat and per protocol analyses | 2 YEARS

SECONDARY OUTCOMES:
Adverse events during treatment | 2 YEARS
  The percentage of patients reporting side effects during treatment and the following days until the evaluation of Hp eradication

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandra General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sugano K, Tack J, Kuipers EJ, Graham DY, El-Omar EM, Miura S, Haruma K, Asaka M, Uemura N, Malfertheiner P; faculty members of Kyoto Global Consensus Conference. Kyoto global consensus report on Helicobacter pylori gastritis. Gut. 2015 Sep;64(9):1353-67. doi: 10.1136/gutjnl-2015-309252. Epub 2015 Jul 17. PMID 26187502
- [Background] Megraud F, Coenen S, Versporten A, Kist M, Lopez-Brea M, Hirschl AM, Andersen LP, Goossens H, Glupczynski Y; Study Group participants. Helicobacter pylori resistance to antibiotics in Europe and its relationship to antibiotic consumption. Gut. 2013 Jan;62(1):34-42. doi: 10.1136/gutjnl-2012-302254. Epub 2012 May 12. PMID 22580412
- [Background] Georgopoulos SD, Xirouchakis E, Martinez-Gonzales B, Zampeli E, Grivas E, Spiliadi C, Sotiropoulou M, Petraki K, Zografos K, Laoudi F, Sgouras D, Mentis A, Kasapidis P, Michopoulos S. Randomized clinical trial comparing ten day concomitant and sequential therapies for Helicobacter pylori eradication in a high clarithromycin resistance area. Eur J Intern Med. 2016 Jul;32:84-90. doi: 10.1016/j.ejim.2016.04.011. Epub 2016 Apr 28. PMID 27134145